CLINICAL TRIAL: NCT01085864
Title: Biomarkers for Diagnosis of Lung Nodules
Acronym: Nodule
Status: Active, not recruiting | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 09-1106.cc
Record Dates: First submitted 2010-03-10; First posted 2010-03-12 (Estimated); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Lung Abscess
Keywords: Lung Nodules; A need exists for non-invasive testing to aid in clinical decision-making for CT scan detected lung nodules of indeterminate etiology.
MeSH Terms: conditions — Lung Abscess

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood specimen, a sputum sample, a urine sample, and an exhaled breath sample.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with lung nodules on CT scan.: Patients with lung nodules on CT scan.

SUMMARY:
A need exists for non-invasive testing to aid in clinical decision-making for Computerized Tomography (CT) scan detected lung nodules of indeterminate etiology. The investigators hypothesize that biomarkers detectable in blood, sputum or urine may be useful for guiding clinical decisions in the setting of CT detected lung nodules to determine which nodules are malignant and which are benign. The investigators also hypothesize that these biomarkers will decrease in concentration to the normal range after successful surgical treatment of malignant lung nodules.

DETAILED DESCRIPTION:
The Biomarkers for Diagnosis of Lung Nodules Study is a prospective study of a cohort of 500 individuals with lung nodules of indeterminate etiology that are identified by CT scans. Either biopsy or repeat CT scans must be clinically indicated to determine the etiology of the nodule. Patients will be asked to allow investigators access to CT scan images and spirometry data, and provide blood, sputum, urine, and exhaled breath samples over the course of the study. Patients will also be asked to allow investigators to access pathology records if a biopsy or surgical excision of the nodule is clinically indicated.

ELIGIBILITY:
Inclusion Criteria:

1. Adult 18-85 years of age
2. Patients referred to pulmonologists, oncologists, or thoracic surgeons for the evaluation of peripheral lung nodules found on CT scan.
3. Repeat CT scans, biopsy or surgical excision are clinically indicated to determine the etiology of the nodule.
4. One or more lung nodules must be between 8 mm and 30 mm in the greatest diameter.
5. Patients must be fully informed of the investigational nature of the procedure and sign an informed consent.

   -

Exclusion Criteria:

1. Lung nodules or masses greater than 30 mm in the greatest dimension.
2. Lung nodules that have solid calcification.
3. Lung nodules or masses with CT evidence of partial or complete obstruction of a lobar bronchus, main stem bronchus or the trachea.
4. No prior cancer with the exception of non-melanoma skin cancer.
5. Life expectancy of < 6 months
6. Any individual who does not give oral and written consent for participation -

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients being evaluated by CT Scan with Lung Nocules
Sampling Method: Probability Sample
Enrollment: 550 (Estimated)
Dates: Start 2010-03-17 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of biomarkers in blood, sputum or urine. | Baseline, 3-6 months, 12 months, 24 months, time of biopsy or surgery (if applicable), and 6 months post surgery (if applicable).
  The primary hypothesis is that biomarkers detectable in blood, sputum, or urine will be useful for guiding clinical decisions in the setting of CT detected lung nodules.

SECONDARY OUTCOMES:
Evaluation of biomarkers after successful surgical treatment of malignant lung nodules. | Within 3 years
  The secondary hypothesis is that these biomarkers will decrease in concentration to the normal range after successful surgical treatment of malignant lung nodules.

CONTACTS AND LOCATIONS:
Overall Officials: York E Miller, M.D., Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States